CLINICAL TRIAL: NCT01466491
Title: Refining Paracervical Block Techniques for Pain Control in First Trimester Surgical Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Planned Parenthood Federation of America (Other)
Responsible Party: Principal Investigator, Paula Bednarek, Assistant Professor, Department of Obstetrics and Gynecology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OHSU SFP 7688
Record Dates: First submitted 2011-11-01; First posted 2011-11-08 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Pain
Keywords: Pain during first-trimester surgical abortion
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 4-site injection (Placebo Comparator): The superior technique of Phase 1 will be compared to a 4-site technique (both techniques will have no wait prior to dilation unless wait was superior in Phase 1).
  Interventions: Drug: Paracervical block technique with lidocaine
- 2-site Injection (Active Comparator): The superior technique of Phase 1 will be compared to a 2-site technique (2 mL injected at the tenaculum site, 18 mL equally distributed between 4 and 8 o'clock) in a randomized fashion (both techniques will have no wait prior to dilation unless wait was superior in Phase 1).
  Interventions: Drug: Paracervical block technique with lidocaine
- 4-Site PCB followed by 3-minute wait (Placebo Comparator): Women will be randomized to receive a 4-site PCB followed by a 3-minute wait (PCB 20/4/3) prior to dilation
  Interventions: Drug: Paracervical block technique with lidocaine
- 4-site PCB followed by no wait (Active Comparator): Women will be randomized to receive a 4-site PCB followed by no wait (PCB 20/4/0).
  Interventions: Drug: Paracervical block technique with lidocaine

INTERVENTIONS:
Drug: Paracervical block technique with lidocaine — The PCB will consist of a total of 20 mL local anesthetic (18 mL of 1% lidocaine buffered with 2 mL sodium bicarbonate) injected with the following technique: 2 mL are injected at the tenaculum site, 12 o'clock, superficially into the cervix. The tenaculum is placed at 12 o'clock. The remaining 18 mL are injected paracervically (vaginal fornices) over sixty seconds. The injection, occurring in either two or four sites, is continuous from superficial to deep (3 cm) to superficial (injecting with insertion and withdrawal). It will be followed with either no wait or a three-minute wait period.

SUMMARY:
The purpose of this study is to determine the level of pain women experience with a surgical abortion and the effect that varying paracervical block techniques might have on that pain. These different techniques involve wait time following the injection as well as the number of sites injected.

DETAILED DESCRIPTION:
The investigators plan to conduct a single-blinded randomized trial of 350 women undergoing elective first-trimester surgical abortion. Subjects will be randomized to two different paracervical block techniques, but both the medications and the amount of medications will remain the same. Subjects will not know to which group they have been randomized as this knowledge may affect how much pain is felt.

Primary Outcome:

Patient reported pain with cervical dilation during first trimester surgical abortion. Pain is measured as mm distance from the left of the 100-mm visual analogue (VAS) scale with the anchors 0 = none, 100 mm = worst imaginable (reflecting magnitude of pain) and recorded immediately after completion of cervical dilation. The 100-mm VAS scale is a well established and validated study instrument.

Secondary Outcomes:

1. Socio-demographic and clinical data: age, race, gravidity, parity, gestational age, prior vaginal delivery, prior abortion, level of menstrual symptoms
2. Pain (VAS scale):

   * anticipated
   * baseline
   * with speculum insertion
   * with placement of the PCB
   * with aspiration
   * 30 min postoperatively
   * intrapersonal pain changes (calculated in analysis)
   * anxiety [baseline] (VAS scale; anchors 0 = none, 100mm = worst imaginable):
   * of pain
   * of surgery
   * satisfaction (VAS scale; anchors 0 = not, 100mm = very satisfied):
   * with pain control
   * overall abortion experience
   * adverse events
   * need for additional intraoperative and/or postoperative pain medication
   * participants' belief if they were in the intervention or control group

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* voluntarily requesting pregnancy termination
* ultrasound-confirmed intrauterine pregnancy up to 10 6/7 weeks gestational age
* generally healthy
* English or Spanish speaking
* able or willing to sign an informed consent and agree to terms of the study

Exclusion Criteria:

* gestational age over 10 6/7 weeks (due to routine use of misoprostol starting at this gestational age at the study sites)
* incomplete abortion
* failed medical abortion
* required or requested IV sedation (prior to randomization)
* patient who declines Ibuprofen, Lorazepam or PCB
* medical contraindication or allergy to any of the study medications
* chronic use of narcotic pain medication or heroin
* significant physical or mental health condition
* adnexal mass or tenderness on pelvic exam consistent with inflammatory disease
* known hepatic disease
* women who, in the opinion of the investigator, are not suitable for the study protocol

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Bednarek, MD MPH, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - Planned Parenthood Columbia Willamette, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4-site Injection | 2-site Injection | 4-Site PCB Followed by 3-minute Wait | 4-site PCB Followed by no Wait
Started | 83 | 83 | 83 | 83
Completed | 83 | 80 | 80 | 83
Not Completed | 0 | 3 | 3 | 0
Not completed — Protocol Violation | 0 | 3 | 2 | 0
Not completed — Missing Data | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4-site Injection | 2-site Injection | 4-Site PCB Followed by 3-minute Wait | 4-site PCB Followed by no Wait | Total
Number analyzed (Participants) | 83 | 80 | 80 | 83 | 326
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 83 | 80 | 80 | 83 | 326
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (5.2) | 25.5 (5.3) | 25.2 (5.2) | 26.4 (5.5) | 25.575 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 80 | 80 | 83 | 326
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 83 | 80 | 80 | 83 | 326

OUTCOME MEASURES:

1. Primary Outcome: Patient Perception of Pain
Description: To determine whether varying paracervical block techniques affect patient perception of pain. Pain is measured as mm distance from the left of the 100-mm visual analogue (VAS) scale with the anchors 0 = none, 100 mm = worst imaginable (reflecting magnitude of pain) and recorded immediately after completion of cervical dilation.
Time Frame: after completion of cervical dilation
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 4-site Injection | 2-site Injection | 4-Site PCB Followed by 3-minute Wait | 4-site PCB Followed by no Wait
Number analyzed (Participants) | 83 | 80 | 80 | 83
mm | 60 (30) | 68 (21) | 56 (32) | 63 (24)

2. Secondary Outcome: Pain Scores Throughout Procedure at Various Time Points
Description: Distance (mm) from the left of the 100 mm Visual Analog Scale (VAS anchors: 0=none, 100 mm= worst imaginable) recorded at various points throughout procedure:
  * prior to medication (baseline)
  * after speculum insertion
  * with placement of PCB
  * with cervical dilation
  * with aspiration
  * 30 minutes post-operatively
Time Frame: up to several hours
Measure: Mean (Standard Error); unit: mm
Arm/Group | 4-site Injection | 2-site Injection | 4-Site PCB Followed by 3-minute Wait | 4-site PCB Followed by no Wait
Number analyzed (Participants) | 83 | 80 | 80 | 83
mm
  Prior to medication (baseline) | 7.65 (1.27) | 4.84 (1.30) | 4.2 (2.5) | 6 (0.9)
  After speculum insertion | 29.35 (2.43) | 27.31 (2.47) | 29.3 (2.7) | 30.3 (2.7)
  With placement of PCB | 58.89 (2.64) | 55.31 (2.69) | 60.0 (2.8) | 58.3 (2.8)
  With cervical dilation | 59.76 (2.84) | 68.41 (2.90) | 55.6 (3.1) | 63.2 (3.1)
  With aspiration | 67.75 (2.52) | 74.05 (2.56) | 72.1 (2.6) | 69.4 (2.5)
  30 minutes post-operatively | 26.27 (2.56) | 22.37 (2.30) | 27.3 (2.6) | 24.2 (2.5)

ADVERSE EVENTS:
Time Frame: During procedure to 30 minutes post-procedure.
Arm/Group | 4-site Injection | 2-site Injection | 4-Site PCB Followed by 3-minute Wait | 4-site PCB Followed by no Wait
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/80 | 0/80 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/80 | 0/80 | 0/83
Other Adverse Events (participants affected / at risk) | 0/83 | 0/80 | 0/80 | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No